CLINICAL TRIAL: NCT03334149
Title: Blood Pressure Monitoring in High Risk Pregnancy to Improve the Detection and Monitoring of Hypertension
Acronym: BUMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: King's College London (Other); Oxford University Hospitals NHS Trust (Other); University of Southampton (Other); University of Birmingham (Other); Barts & The London NHS Trust (Other); City, University of London (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 224978
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy, High Risk; Pre-Eclampsia; Hypertension; Hypertension, Pregnancy-Induced
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Intervention Model Description: Note Women in BUMP 1 will transfer to BUMP 2 if they develop hypertension. Women in BUMP 2 can be randomised de novo or join from BUMP 1 maintaining their original randomisation. The enrolment number below therefore includes BUMP 1 (2262) plus BUMP 2 (512). Permission was granted by the ethics committee to continue recruitment passed the original sample size until the original planned end of recruitment date.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Monitoring of Blood Pressure (Experimental): BUMP 1: using a validated home blood pressure monitor at least 3 times a week to record blood pressure BUMP 2: using a validated home blood pressure monitor daily to record blood pressure Women in the intervention groups will be encouraged to use a simple mobile tele monitoring system.
  Interventions: Other: Self-Monitoring of Blood Pressure
- Usual Care (No Intervention): Women randomised to usual care will continue to have all their BP monitoring completed by the clinical team at their antenatal assessments.

INTERVENTIONS:
Other: Self-Monitoring of Blood Pressure — BUMP 1: Women randomised to the self-monitoring arm will be asked to measure blood pressures at least three times a week. They will perform two readings with a one minute interval and will be asked to act on the second reading if it falls outside their normal range thresholds described in their instructions, and aided by the tele monitoring system.
  BUMP 2: Women randomised to the self-monitoring arm will be asked to measure blood pressures daily. They will perform two readings with a one minute interval and will be asked to act on the second reading if it falls outside their normal range thresholds described in their instructions, aided by a tele monitoring system.
  Arms: Self-Monitoring of Blood Pressure

SUMMARY:
Raised blood pressure is a common problem in pregnancy. Raised blood pressure and pre-eclampsia affect about one in ten women and are a major cause of death and premature birth in the United Kingdom and worldwide.

Many women have expressed an interest in monitoring their own blood pressure in between antenatal visits but there has been very little research to guide this. The investigators would like to know if the diagnosis and subsequent care of women with raised blood pressure can be improved if women were able to monitor their own blood pressure safely at home. This work will test whether optimising the diagnosis, monitoring and management of raised BP during pregnancy through self-monitoring of BP is effective, acceptable and cost-effective compared to usual care.

The research team have being working with pregnant women, doctors and midwives to develop a simple and accurate method of self-monitoring of blood pressure in pregnancy.

This randomised controlled trial will:

1. Compare self-monitoring with usual care in women at higher risk of hypertension in pregnancy and assess if self-monitoring can identify raised blood pressure earlier.
2. Compare self-monitoring with usual care for women with high blood pressure in pregnancy to see if it leads to lower blood pressure.
3. Assess if self-monitoring is cost-effective.

Pregnant women who chose to take part in these studies will be randomised to either usual care or asked to monitor their own blood pressure during their pregnancy in addition to their usual antenatal care.

DETAILED DESCRIPTION:
BUMP 1 will randomise 2262 women at higher risk of hypertension in pregnancy into usual care or self-monitoring.

BUMP 2 will randomise 512 women with hypertension in pregnancy (including chronic hypertension) into usual care or self-monitoring. Women in BUMP 1 will move into BUMP 2 if they develop hypertension.

Women will be recruited at approximately 15 hospitals in England over approximately 24 months.

Women will be recruited from 20 weeks (BUMP 1) or early pregnancy(BUMP 2) and followed up until 2 months after birth.

ELIGIBILITY:
BUMP 1

Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Pregnant woman, aged 18 years or above between 16+0 to 24+0 weeks
* Able and willing to comply with trial requirements
* Willing to allow her general practitioner and consultant, if appropriate, to be notified of participation in the trial
* At higher risk for hypertension in pregnancy / pre-eclampsia defined as one or more of the following risk factors:
* Age 40 years or older
* Nulliparity
* Pregnancy interval of more than 10 years
* Family history of pre-eclampsia
* Previous history of pre-eclampsia or gestational hypertension
* Body mass index 30 kg/m2 or above at booking
* Chronic kidney disease
* Twin pregnancy
* Diabetes (Type 1&2)
* Autoimmune Disease (eg systemic lupus erythematosis or antiphospholipid disease)

Exclusion Criteria:

* Chronic Hypertension

BUMP 2:

Inclusion Criteria:

• Women developing pregnancy hypertension previously randomised in BUMP 1 (regardless of gestation).

OR

* Women with chronic hypertension (defined as sustained systolic BP≥140 mmHg and/or diastolic BP≥90 mmHg, present at booking or before 20 weeks' gestation, or receiving treatment outside pregnancy and/or at time of referral).
* Recruited up to 37+0 weeks' gestation.

OR

* Women with hypertension after 20 weeks' gestation (defined as sustained systolic BP≥140 mmHg and/or diastolic BP≥90 mmHg).
* Recruited at 20+0 to 37+0 weeks' gestation.

AND

* Participant is willing and able to give informed consent for participation in the trial.
* Woman aged 18 years or above.
* Willing to allow her general practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion criteria:

Anticipated inpatient admission considered likely to lead to imminent delivery (within the next 48 hours)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Women
Enrollment: 3042 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Time from recruitment to diagnosis of raised blood pressure | From study entry to delivery i.e. up to approximately 25 weeks from recruitment
  Difference between groups in time from recruitment to recording of raised blood pressure by health care professional.
Mean systolic blood pressure | From study entry to delivery i.e. up to 40 weeks
  Difference in mean systolic blood pressure between usual care and self-monitoring group.

SECONDARY OUTCOMES:
Severe hypertension | From study entry to delivery i.e. up to 40 weeks
  Difference between usual care and self-monitoring group in severe hypertension (systolic BP ≥160mmHg and/or or diastolic BP ≥110mmHg) (BUMP 1 and BUMP 2)
Serious maternal complications | From study entry to delivery i.e. up to 40 weeks
  Difference between usual care and self-monitoring group in serious maternal complications (pre-eclampsia, placental abruption, transient ischemic attack or stroke, pulmonary oedema, renal failure, blood transfusion), death (BUMP 1 and BUMP 2)
Onset of labour | At delivery
  Difference between usual care and self-monitoring group in onset of labour (BUMP 1 and BUMP 2)
Assessment of quality of life differences between arms | From study entry to 30 weeks of pregnancy, or from study entry to 2 weeks following study entry if randomised after 30 weeks pregnancy
  Difference between usual care and self-monitoring group in change in quality of life (measured using the EQ-5D-5L) (BUMP 1 and BUMP 2)
Assessment of quality of life differences between arms | From study entry to 8 weeks postpartum i.e. up to 48 weeks
  Difference between usual care and self-monitoring group in change in quality of life (measured using the EQ-5D-5L (BUMP 1 and BUMP 2)
Stillbirth | At delivery
  Difference between usual care and self-monitoring group in number of stillbirths (BUMP 1 and BUMP 2)
Early neonatal deaths | From delivery up to 28 days postpartum i.e. up to 4 weeks
  Difference between usual care and self-monitoring group in number of early neonatal deaths (BUMP 1 BUMP 2)
Gestation at delivery | At delivery
  Difference between usual care and self-monitoring group in gestation at delivery (BUMP 1 and BUMP 2)
Mode of delivery | At delivery
  Difference between usual care and self-monitoring group in mode of delivery (BUMP 1 and BUMP 2)
Birth weight including centile | At delivery
  Difference between usual care and self-monitoring group in birth weight of the baby including centile (BUMP 1 and BUMP 2)
Small for gestational age infants | At delivery
  Difference between usual care and self-monitoring group in number of small for gestational age infants (<10th and <3rd centile) (BUMP 1 and BUMP 2)
Neonatal unit admissions | From delivery up to 28 days postpartum i.e. up to 4 weeks
  Difference between usual care and self-monitoring group in number of neonatal unit admissions including length of stay (BUMP 1 and BUMP 2)
Health behaviours | From study entry to 30 weeks of pregnancy, or from study entry to 2 weeks following study entry if randomised after 30 weeks pregnancy.
  Difference between usual care and self-monitoring group in change in health behaviours (questionnaire) (BUMP 1 and BUMP 2)
Health behaviours | From study entry to 8 weeks postnatal i.e. up to 48 weeks
  Difference between usual care and self-monitoring group in change in health behaviours (questionnaire) (BUMP 1 and BUMP 2)
Fidelity to monitoring schedule | From study entry to delivery i.e. up to 48 weeks
  Difference between usual care and self-monitoring group in fidelity to monitoring schedule (BUMP 1 and BUMP 2)
STAI-6 short form anxiety questionnaire | From study entry to 30 weeks of pregnancy, or from study entry to 2 weeks following study entry if randomised after 30 weeks pregnancy.
  Difference between usual care and self-monitoring group in change in State trait anxiety inventory short form anxiety questionnaire (STAI-6 ) (BUMP 1 and BUMP 2)
STAI-6 short form anxiety questionnaire | From study entry to 8 weeks postnatal i.e. up to 48 weeks
  Difference between usual care and self-monitoring group in change in STAI-6 short form anxiety questionnaire (BUMP 1 and BUMP 2)
Health service costs | From study entry to delivery i.e. up to 40 weeks
  Difference between usual care and self-monitoring group in health service costs. (BUMP 1 and BUMP 2)
Cost per quality-adjusted life year gained over trial period | From study entry to delivery i.e. up to 40 weeks
  Difference between usual care and self-monitoring group in cost per quality-adjusted life year gained over trial period (BUMP 1 and BUMP 2)
Qualitative | From study entry to 8 weeks postpartum i.e. up to 48 weeks
  Qualitative data gathered from participating women and healthcare professionals (BUMP 1 and BUMP 2)
Mean diastolic blood pressure | From study entry to delivery i.e. up to 40 weeks
  Difference between usual care and self-monitoring group in mean diastolic blood pressure (BUMP 2)
Mean area under the blood pressure over time curve | From study entry to delivery i.e. up to 40 weeks
  Difference between usual care and self-monitoring group in mean area under the blood pressure curve (BUMP 2)
Mean proportion of readings above 140mmHg | From study entry to delivery i.e. up to 40 weeks
  Difference between usual care and self-monitoring group in mean proportion of readings above 140mmHg (BUMP 2)
Adherence to medication | From study entry to 30 weeks of pregnancy, or from study entry to 2 weeks following study entry if randomised after 30 weeks pregnancy.
  Difference between usual care and self-monitoring group in change in adherence to medication (MARS) (BUMP 2)
Adherence to medication | From study entry to 8 weeks postnatal i.e. up to 48 weeks
  Difference between usual care and self-monitoring group in change in adherence to medication (MARS) (BUMP 2)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J McManus, PhD MBBS, Principal Investigator — University of Oxford
Locations (13):
- United Kingdom (13):
  - Buckinghamshire Healthcare NHS Trust, Aylesbury
  - Birmingham Women's and Children's Hospital NHS Foundation Trust, Birmingham
  - Croydon Health Services NHS Trust, London
  - Barts Health NHS Trust, London
  - Kingston Hospital NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - The Royal Berkshire NHS Foundation Trust, Reading
  - The Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Data are available from the authors upon reasonable request and with permission of the University of Oxford. Use of data will require approval by an independent review committee identified for this purpose and investigators requesting data will need to provide a written protocol including analysis plan and sign a data sharing/access agreement. Requests for Data Sharing should be directed to information.guardian@phc.ox.ac.uk.
Supporting Information: Study Protocol, SAP
Time Frame: from 31st May 2023
Access Criteria: Use of data will require approval by an independent review committee identified for this purpose and investigators requesting data will need to provide a written protocol including analysis plan and sign a data sharing/access agreement.

REFERENCES:
- [Background] Dougall G, Franssen M, Tucker KL, Yu LM, Hinton L, Rivero-Arias O, Abel L, Allen J, Band RJ, Chisholm A, Crawford C, Green M, Greenfield S, Hodgkinson J, Leeson P, McCourt C, MacKillop L, Nickless A, Sandall J, Santos M, Tarassenko L, Velardo C, Wilson H, Yardley L, Chappell L, McManus RJ. Blood pressure monitoring in high-risk pregnancy to improve the detection and monitoring of hypertension (the BUMP 1 and 2 trials): protocol for two linked randomised controlled trials. BMJ Open. 2020 Jan 23;10(1):e034593. doi: 10.1136/bmjopen-2019-034593. PMID 31980512
- [Result] Tucker KL, Mort S, Yu LM, Campbell H, Rivero-Arias O, Wilson HM, Allen J, Band R, Chisholm A, Crawford C, Dougall G, Engonidou L, Franssen M, Green M, Greenfield S, Hinton L, Hodgkinson J, Lavallee L, Leeson P, McCourt C, Mackillop L, Sandall J, Santos M, Tarassenko L, Velardo C, Yardley L, Chappell LC, McManus RJ; BUMP Investigators. Effect of Self-monitoring of Blood Pressure on Diagnosis of Hypertension During Higher-Risk Pregnancy: The BUMP 1 Randomized Clinical Trial. JAMA. 2022 May 3;327(17):1656-1665. doi: 10.1001/jama.2022.4712. PMID 35503346
- [Result] Chappell LC, Tucker KL, Galal U, Yu LM, Campbell H, Rivero-Arias O, Allen J, Band R, Chisholm A, Crawford C, Dougall G, Engonidou L, Franssen M, Green M, Greenfield S, Hinton L, Hodgkinson J, Lavallee L, Leeson P, McCourt C, Mackillop L, Sandall J, Santos M, Tarassenko L, Velardo C, Wilson H, Yardley L, McManus RJ; BUMP 2 Investigators. Effect of Self-monitoring of Blood Pressure on Blood Pressure Control in Pregnant Individuals With Chronic or Gestational Hypertension: The BUMP 2 Randomized Clinical Trial. JAMA. 2022 May 3;327(17):1666-1678. doi: 10.1001/jama.2022.4726. PMID 35503345
- [Derived] Campbell HE, Chappell LC, McManus RJ, Tucker KL, Crawford C, Green M, Rivero-Arias O. Detection and Control of Pregnancy Hypertension Using Self-Monitoring of Blood Pressure With Automated Telemonitoring: Cost Analyses of the BUMP Randomized Trials. Hypertension. 2024 Apr;81(4):887-896. doi: 10.1161/HYPERTENSIONAHA.123.22059. Epub 2024 Jan 23. PMID 38258566
- [Derived] Hinton L, Hodgkinson J, Tucker KL, Rozmovits L, Chappell L, Greenfield S, McCourt C, Sandall J, McManus RJ. Exploring the potential for introducing home monitoring of blood pressure during pregnancy into maternity care: current views and experiences of staff-a qualitative study. BMJ Open. 2020 Dec 1;10(12):e037874. doi: 10.1136/bmjopen-2020-037874. PMID 33262186
- [Derived] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394